CLINICAL TRIAL: NCT05751915
Title: Magnetocardiography as a Noninvasive Diagnostic Strategy for Identifying Coronary Allograft Vasculopathy
Acronym: M-CAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Genetesis Inc. (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 10007
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Coronary Allograft Vasculopathy (CAV)
Keywords: Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- PET CAV 0: Normal perfusion with normal global stress (> 1.7 mL/min/g)
  Interventions: Device: CardioFlux
- PET CAV 1: Normal perfusion with abnormal global stress MBF (<1.7 mL/min/g and ejection fraction >45%) OR Single vessel perfusion defect with normal global stress MBF.
  Interventions: Device: CardioFlux
- PET CAV 2/3: Normal perfusion with abnormal global stress MBF (<1.7 mL/min/g) and ejection fraction < 45% OR Single vessel perfusion defect with abnormal global stress MBF (<1.7 mL/min/g) OR Multivessel perfusion defects v
  Interventions: Device: CardioFlux

INTERVENTIONS:
Device: CardioFlux — CardioFlux MCG is a process that observes incremental changes in the heart's electrical activity by the magnetic fields generated by these currents. These magnetic fields have been used for decades via electrocardiogram to help diagnose and treat both acute and chronic cardiac pathology. The CardioFlux device reaches the potential of this phenomenon by sensing a complete magnetic field map. It is equipped with a magnetic shielding chamber and can attenuate magnetic field noise by a factor of nearly 1500 which maximizes signal to noise ratio. CardioFlux is an easy to operate, noninvasive modality that can detect the presence of ischemic cardiac tissue in symptomatic patients in a less than 5-minute scan. The device uses the proprietary software called Faraday which processes MCG scans, create diagnostic functional images, and run analytics.

SUMMARY:
Purpose: To show early feasibility of magnetocardiography (MCG) to identify coronary Cardiac positron emission tomography (PET) is the preferred non-invasive tests to assess for CAV and incorporation of quantitative myocardial blood flow (MBF) assessment improves diagnostic accuracy. Based on ISHLT criteria, the following have been proposed for diagnosis of CAV by PET:

DETAILED DESCRIPTION:
Diagnosing CAV by PET with quantitative myocardial blood flow (MBF) 3 PET CAV 0: Normal perfusion with normal global stress (> 1.7 mL/min/g)

PET CAV 1: Normal perfusion with abnormal global stress MBF (<1.7 mL/min/g and ejection fraction >45%) OR Single vessel perfusion defect with normal global stress MBF.

PET CAV 2/3: Normal perfusion with abnormal global stress MBF (<1.7 mL/min/g) and ejection fraction < 45% OR Single vessel perfusion defect with abnormal global stress MBF (<1.7 mL/min/g) OR Multivessel perfusion defects

With these diagnostic criteria, PET CAV 0 has been shown to have a high negative predictive value for moderate to severe CAV by invasive coronary angiography, and PET CAV 2/3 has been shown to have a high positive predictive value for moderate to severe CAV and is associated with adverse events.

This study further examines the feasibility of MCG in identifying CAV in adult heart transplant recipients and compares those results to the current non-invasive standard using PET CAV scores. This will help determine whether MCG is a potential test for regular surveillance of CAV in transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of enrollment

Willing to provide written informed consent

Completed cardiac PET within the last 2 weeks

No changes to medication or intervention since the PET was completed

Exclusion Criteria:

* Patients unable to fit into device

Patients unable to lie supine for 5 minutes

Patients with implanted ferromagnetic objects above the costal margin of the rib cage (implanted pacemakers, cardioverter/defibrillators, infusion pumps, and/or neuro stimulators).

NOTE: Sternotomy wires stents are acceptable

Implanted pacemakers or cardioverter/defibrillators

Implanted infusion pumps and/or neuro stimulators

Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant recipients are susceptible to developing coronary allograft vasculopathy (CAV), a disease that causes blockages in the arteries of the transplanted heart. CAV often progresses without symptoms, and transplant recipients undergo regular surveillance to detect CAV. Current tests used to detect CAV, such as invasive coronary angiography (ICA) and intravascular ultrasound (US) have clear limitations; in addition to being invasive with risk of complications, they are also expensive, time consuming, and require iodinated contrast, a concern in a population with high rates of kidney dysfunction. In addition, these tests may not be able to detect CAV in its early stages. Additionally, the diagnosis of CAV remains a challenge as angiography, the standard method for detecting focal plaques, lacks sensitivity in detecting CAV, and intravascular ultrasonography, a more sensitive method, lacks the ability to evaluate the entirety of the coronary arteries.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
To compare the performance (diagnostic capabilities) of magnetocardiography in the diagnosis of coronary vasculopathy (CAV) as compared to PET as the currently accepted gold standard non-invasive tool. | 6 months
  Ability of MCG to identify CAV 0 in heart transplant patients as measured by sensitivity, specificity, positive predictive value, and negative predictive value.

SECONDARY OUTCOMES:
To determine whether MCG is able to differentiate between CAV 0, 1, and 2/3, and to correlate with absolute stress myocardial blood flow, global CFR (Coronary flow reserve), and LVEF (Left ventricular ejection fraction), as measured by cardiac PET | 6 months
  Differentiation between CAV 0, 1, and 2/3
  Correlation of MCG with absolute stress myocardial blood flow
  Correlation of MCG with global CFR
  Correlation of MCG with LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cremer, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No